CLINICAL TRIAL: NCT03177213
Title: Serum IL-21 Levels in Patients With Pemphigus Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Kassim, AssiutU, Assiut University
Other Study IDs: IL-21PV
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pemphigus vulgaris patients: 20 pemphigus vulgaris patients will be included in the study, either newly diagnosed or recurrent. Patients will be recruited on admission from Dermatology department and Outpatient Clinic, Assiut University Hospitals
- Healthy controls: 10 healthy age and sex matched subjects will be included as controls.

SUMMARY:
Pemphigus is severe antigen derived autoimmune bullous skin disorder, the word pemphigus is derived from the Greek word" pemphix " which means blister . Two main clinical variants are known pemphigus vulgaris (PV), and pemphigu foliaceus (PF). (Zenzo .et al., 2015).

DETAILED DESCRIPTION:
Clinically, there are localized or generalized flaccid bullae that quickly transform into post-bullous erosions and crusts , PV patients characteristically develop oral lesions with buccal and/or gingival persisting erosions (mucosal dominant PV) which several weeks or months later may also spread to the epidermis (mucocutaneous PV). PF is characterized by widespread cutaneous fragile bullae which rapidly rupture, resulting in erosions, crusting, and scaling. In contrast to PV, the mucosa is usually not involved in PV. (Zenzo .et al .,2015).

Pathophysiologically, the underlying intraepithelial blister formation is caused by IgG autoantibodies against the desmosomal adhesion proteins, desmoglein 3 and/or desmoglein 1, on epidermal keratinocytes. ( Amagai .et al .,1991) In PV the antigen is desmoglein 3 which is presented in lower epidermis and is expressed more strongly in buccal mucosa than in the skin ,in contrast to PF which its antigen is desmoglein 1 which is expressed in the skin throughout the epidermis and weakly expressed in the mucous membranes . ( Kneisel and Hertl. .,2011).

T cells play a crucial role in the pathogenesis of pemphigus vulgaris , The interaction of T and B cells critically modulates the development of pemphigus vulgaris. (Amber. et al., 2013 ; Zhu, et al.,2012).

Because B-cell activation and antibody production classically necessitate the involvement of CD4+ T cells, Dsg-reactive T cells were capable of recognizing multiple epitopes of the extracellular domain of Dsg and helping B cells to produce a specific antibody. Dsg3-reactive T-cell clones were able to commit polyclonal naive B cells to produce pathogenic anti-Dsg3 antibody and induce the PV phenotype. (Hertl . et al., 1998) Follicular T helper cells (Tfh) are a recently discovered group of CD4+ Th cells with intrinsic differences from Th1, Th2 and Th17 cells. Localized in B-cell follicles of secondary lymphoid tissues, The major function of Tfh cells appears to help B-cell activation and antibody production during humoral immune responses. The Tfh cells express high levels of IL-21, which was demonstrated to be important for the generation of Tfh cells and that responsiveness of Tfh cells to IL-21 drives the formation of the autoimmune reaction, and it clearly impacted on the amount of antibody production.( Gomez. et al.,2011 ; Vogelzang . et al.,2008) Nowadays, finding a promising treatment for pemphigus remains a serious challenge. Various treatments are currently recommended to treat this disease, but they rarely lead to complete and durable remission. Regulatory cells appear to have a critical role in numerous autoimmune diseases, so it is possible that control of these cells may induce remission. (Cholera and Chainani .,2016)

ELIGIBILITY:
Inclusion Criteria:

* 20 pemphigus vulgaris patients
* healthy age and sex matched

Exclusion Criteria:

* - Patients with a history of topical or systemic treatment (corticosteroids, intralesional steroid injection, immunosuppressive therapy, anticonvulsants and anticancer medications, within 4 weeks of the study.
* Patients receiving phototherapy within 6 months of the study .
* Patients with a history of diabetes mellitus, anemia, thyroid or parathyroid disorders, chronic liver or renal diseases, or atopy .
* Patients with known autoimmune diseases or cancer.
* Pregnant or lactating women were also excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 20 pemphigus vulgaris patients will be included in the study, either newly diagnosed or recurrent. Patients will be recruited on admission from Dermatology department and Outpatient Clinic, Assiut University Hospitals. 10 healthy age and sex matched subjects will be included as controls.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
serum IL-21 | 2 months
  serum IL-21 level

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu H, Chen Y, Zhou Y, Wang Y, Zheng J, Pan M. Cognate Th2-B cell interaction is essential for the autoantibody production in pemphigus vulgaris. J Clin Immunol. 2012 Feb;32(1):114-23. doi: 10.1007/s10875-011-9597-4. Epub 2011 Oct 19. PMID 22009001
- [Result] Amber KT, Staropoli P, Shiman MI, Elgart GW, Hertl M. Autoreactive T cells in the immune pathogenesis of pemphigus vulgaris. Exp Dermatol. 2013 Nov;22(11):699-704. doi: 10.1111/exd.12229. PMID 24433179
- [Result] Amagai M, Klaus-Kovtun V, Stanley JR. Autoantibodies against a novel epithelial cadherin in pemphigus vulgaris, a disease of cell adhesion. Cell. 1991 Nov 29;67(5):869-77. doi: 10.1016/0092-8674(91)90360-b. PMID 1720352
- [Result] Cholera M, Chainani-Wu N. Management of Pemphigus Vulgaris. Adv Ther. 2016 Jun;33(6):910-58. doi: 10.1007/s12325-016-0343-4. Epub 2016 Jun 10. PMID 27287854
- [Result] Di Zenzo G, Amber KT, Sayar BS, Muller EJ, Borradori L. Immune response in pemphigus and beyond: progresses and emerging concepts. Semin Immunopathol. 2016 Jan;38(1):57-74. doi: 10.1007/s00281-015-0541-1. Epub 2015 Nov 23. PMID 26597100
- [Result] Gomez-Martin D, Diaz-Zamudio M, Romo-Tena J, Ibarra-Sanchez MJ, Alcocer-Varela J. Follicular helper T cells poise immune responses to the development of autoimmune pathology. Autoimmun Rev. 2011 Apr;10(6):325-30. doi: 10.1016/j.autrev.2010.11.007. Epub 2010 Dec 15. PMID 21167320
- [Result] Hertl M, Amagai M, Sundaram H, Stanley J, Ishii K, Katz SI. Recognition of desmoglein 3 by autoreactive T cells in pemphigus vulgaris patients and normals. J Invest Dermatol. 1998 Jan;110(1):62-6. doi: 10.1046/j.1523-1747.1998.00086.x. PMID 9424089
- [Result] Kneisel A, Hertl M. Autoimmune bullous skin diseases. Part 1: Clinical manifestations. J Dtsch Dermatol Ges. 2011 Oct;9(10):844-56; quiz 857. doi: 10.1111/j.1610-0387.2011.07793.x. English, German. PMID 21955378
- [Result] Kneisel A, Hertl M. Autoimmune bullous skin diseases. Part 2: diagnosis and therapy. J Dtsch Dermatol Ges. 2011 Nov;9(11):927-47. doi: 10.1111/j.1610-0387.2011.07809.x. English, German. PMID 22026362
- [Result] Rosenbach M, Murrell DF, Bystryn JC, Dulay S, Dick S, Fakharzadeh S, Hall R, Korman NJ, Lin J, Okawa J, Pandya AG, Payne AS, Rose M, Rubenstein D, Woodley D, Vittorio C, Werth BB, Williams EA, Taylor L, Troxel AB, Werth VP. Reliability and convergent validity of two outcome instruments for pemphigus. J Invest Dermatol. 2009 Oct;129(10):2404-10. doi: 10.1038/jid.2009.72. Epub 2009 Apr 9. PMID 19357707
- [Result] Vogelzang A, McGuire HM, Yu D, Sprent J, Mackay CR, King C. A fundamental role for interleukin-21 in the generation of T follicular helper cells. Immunity. 2008 Jul 18;29(1):127-37. doi: 10.1016/j.immuni.2008.06.001. Epub 2008 Jul 3. PMID 18602282